CLINICAL TRIAL: NCT05632341
Title: GCWB1176 8 Weeks, Multi -Tube, Randomized Assignment, Double -Eye, Placebo Control Human Application Test for Evaluating the Effectiveness and Safety of the Immune Function
Brief Title: GCWB1176 Evaluates the Effectiveness and Safety of Immune Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Wellbeing (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GCWB110
Record Dates: First submitted 2022-11-11; First posted 2022-11-30 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-11

CONDITIONS: Immune Function
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GCWB1176 (Experimental): 1 capsule once a day
  Interventions: Dietary Supplement: Lactococcus lactis
- Placebo (Active Comparator): 1 capsule once a day
  Interventions: Other: maltodextrin

INTERVENTIONS:
Dietary Supplement: Lactococcus lactis — 1 capsule once a day
  Arms: GCWB1176
Other: maltodextrin — 1 capsule once a day
  Arms: Placebo

SUMMARY:
This human application test was planned to evaluate the effectiveness and safety of immunodefinition compared to the placebo when the GCWB1176 was consumed for those whose white blood cell level was normal or somewhat decreased.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of screening, 19 or 75 years
2. A person with a peripheral blood leukocyte level measured in Visit 1, 3x10^3 cells/μl or more, 8x10^3 cells/μl
3. Those who are more than one of the following standards

   * Those who had more than twice within one year of visiting 1 year.

     * {Common cold, acute tonsillitis, acute pharyngitis, acute laryngitis, acute rhinitis, etc.

       * Those who have stomatitis more than twice within 1 year of visit

         * Those who had Herpes Zoster infection within 1 year of visit
4. Those with a stress awareness scale (PSS) 16 or more
5. A person who agrees to participate in this human application test before the start of the human test and writes a written consent form

Exclusion Criteria:

1. Those who are currently treating drugs due to underlying disease, etc.
2. Hypertension patients (systolic blood pressure 140 mmHg or higher or dichotomous blood pressure 90 mmHg or higher, human application test target 10 minutes stabilized)
3. Patients with diabetes with an fasting blood sugar at least 126 mg/dL or administering urine disease (oral blood sugar, insulin, etc.)
4. Those who are 0.1 UIU/mL or less, or 10 UIU/mL or more
5. Those who have vaccinated vaccines (influenza, corona, shingles that can affect immunity) within 3 months of visiting 1
6. A disease that can affect immune responses such as adult -like and rhinitis
7. AST (GOT) or ALT (GPT) is three times more than the normal upper limit of the embodiment
8. Those who are 1.5 times more than the normal upper limit of Creatinine
9. Those who administered steroids, antibiotics, immunosuppressants, and gastric acid inhibitors within 1 month of visit.
10. Visit 1 person who consumes vitamins, health functional foods that can affect immunity within 2 weeks of visiting
11. A person who has administered or consumed lactic acid bacteria products (4 or more times a week) within 2 weeks of visiting within 2 weeks of visit.
12. Those who complain of severe gastrointestinal symptoms such as heartburn and indigestion
13. Those who are pregnant or have a planning plan for lactation or this human application period
14. Those who have participated in other interventional clinical trials (including human application test) within 8 weeks of visit, or plan to participate in other interventional clinical trials (including human application tests) after the beginning of this human application test
15. Those who are sensitive or allergic to food ingredients for this human application
16. Those who have a BMI (body mass index) of 30 kg/m2 or more
17. A person who consumed alcohol within 1 month (30 days) based on 1 visit (man> 210 g/week, woman> 140 g/week)
18. Those who judge that the test person is inadequate for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change amoust of NK Cell Activity | week 0, 4 and 8
  The comparison of the military comparison for the change before and after the intake of NK CELL Activity is analyzed using the PAIRED T-TEST, and the degree of change between the test group and the control at at each point is Two Sample T-Test or Wilcoxon Rank Sum Test It is conducted to evaluate whether there is a statistically significant difference.

SECONDARY OUTCOMES:
Change amoust of Cytokine analysis (IFN-γ, TNF-α, IL-4, IL-10, IL-12) | week -2, 0, 4 and 8
  The comparison of the military in the before and after consumption is analyzed using the PAIIRED T-TEST, and the degree of change between the test group and the control group at each time is performed by performing the two sample T-test or the Wilcoxon Rank Sum Test according to whether the normality is satisfied. Evaluate if there is a significant difference.
Change amoust of WBC Count analysis | week -2, 0, 4 and 8
  The comparison of the military in the before and after consumption is analyzed using the PAIIRED T-TEST, and the degree of change between the test group and the control group at each time is performed by performing the two sample T-test or the Wilcoxon Rank Sum Test according to whether the normality is satisfied. Evaluate if there is a significant difference.
Change amoust of FSS Count analysis | week -2, 0, 4 and 8
  The comparison of the military in the before and after consumption is analyzed using the PAIIRED T-TEST, and the degree of change between the test group and the control group at each time is performed by performing the two sample T-test or the Wilcoxon Rank Sum Test according to whether the normality is satisfied. Evaluate if there is a significant difference.
Change amoust of upper respiratory infection analysis | week -2, 0, 4 and 8
  The comparison of the military in the before and after consumption is analyzed using the PAIIRED T-TEST, and the degree of change between the test group and the control group at each time is performed by performing the two sample T-test or the Wilcoxon Rank Sum Test according to whether the normality is satisfied. Evaluate if there is a significant difference.
  If there is a statistically significant difference between the military and clinically significantly significantly significant differences in demographic and lifestyle surveys, ANCOVA can be carried out as a covenant.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul St. Mary's Hospital, College of Medicine, Seoul
  - St. Vincent's Hospital, College of Medicine, Suwon